CLINICAL TRIAL: NCT02945358
Title: Assessment of OHIR Score to Predict a Prolonged Intensive Care Unit Stay for Adult Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: Assessment of OHIR Score to Predict a Prolonged Intensive Care Unit Stay
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Other Study IDs: HE581287
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: ICU Stay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prolonged ICU stay: Group 1: adult cardiac surgery with cardiopulmonary pump with prolonged ICU stay Group 2: adult cardiac surgery with cardiopulmonary pump with non-prolonged ICU stay
  Interventions: Procedure: adult cardiac surgery with cardiopulmonary pump

INTERVENTIONS:
Procedure: adult cardiac surgery with cardiopulmonary pump — Open-heart surgery both coronary artery bypass graft (CABG) and valve surgery

SUMMARY:
A prolonged stay in intensive care unit (ICU) after cardiac surgery with cardiopulmonary bypass increases not only cost of patient care but also morbidity and mortality of patients. The ability to predict which patient has the tendency to have a prolonged ICU stay would help in patient and resource management of the hospital. There are many predictive models aiming at identifying patient at risk of prolonged ICU stay after cardiac surgery with cardiopulmonary bypass but almost all involve the preoperative assessment for proper resource management with one model, Open-Heart Intraoperative Risk (OHIR) Scoring concerning intraoperative manipulatable risk factors to improve anesthetic care and patient outcome. The OHIR model comprises 6 risk factors, 5 of which can be managed intraoperatively, with total score of 7 and a score of ≥ 3 indicating a likely prolonged ICU stay. The objective of this study was to re-validate the performance of OHIR score in the recent context.

DETAILED DESCRIPTION:
This will be a retrospective, observational, analytical study. The study protocol was approved by the Human Research Ethics Committee, Khon Kaen University (HE581287).

The investigators will review all eligible medical records at Srinagarind Hospital and Queen Sirikit Heart Center of the Northeast, Khon Kaen University during January 2013 and December 2014. The extracted data consist of patient's clinical data and all risk factors in the OHIR score. The investigators will apply the OHIR scoring to the data to assess its performance. The investigators will use the same criteria for a prolonged ICU stay as in the previous study, i.e. a stay longer that the median.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-75 undergoing cardiac surgery, both CABG and valvular surgery, with the use of cardiopulmonary bypass.

Exclusion Criteria:

* patients having emergency surgery; receiving special devices such as intra-aortic balloon pump or extracorporeal membrane oxygenation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing open-heart surgery both CABG and valve surgery with cardiopulmonary pump
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Intensive care stay | through study completion, an average of 1 week
  number of hours admitted in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
Locations (2):
- Thailand (2):
  - Queen Sirikit Heart Center, Khon Kaen, Changwat Khon Kaen
  - Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen, Changwat Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Williams TA, Ho KM, Dobb GJ, Finn JC, Knuiman M, Webb SA; Royal Perth Hospital ICU Data Linkage Group. Effect of length of stay in intensive care unit on hospital and long-term mortality of critically ill adult patients. Br J Anaesth. 2010 Apr;104(4):459-64. doi: 10.1093/bja/aeq025. Epub 2010 Feb 25. PMID 20185517
- [Result] Hein OV, Birnbaum J, Wernecke K, England M, Konertz W, Spies C. Prolonged intensive care unit stay in cardiac surgery: risk factors and long-term-survival. Ann Thorac Surg. 2006 Mar;81(3):880-5. doi: 10.1016/j.athoracsur.2005.09.077. PMID 16488688
- [Result] Nakasuji M, Matsushita M, Asada A. Risk factors for prolonged ICU stay in patients following coronary artery bypass grafting with a long duration of cardiopulmonary bypass. J Anesth. 2005;19(2):118-23. doi: 10.1007/s00540-005-0301-9. PMID 15875128
- [Result] Gruenberg DA, Shelton W, Rose SL, Rutter AE, Socaris S, McGee G. Factors influencing length of stay in the intensive care unit. Am J Crit Care. 2006 Sep;15(5):502-9. PMID 16926372
- [Result] Almashrafi A, Alsabti H, Mukaddirov M, Balan B, Aylin P. Factors associated with prolonged length of stay following cardiac surgery in a major referral hospital in Oman: a retrospective observational study. BMJ Open. 2016 Jun 8;6(6):e010764. doi: 10.1136/bmjopen-2015-010764. PMID 27279475
- [Result] Almashrafi A, Elmontsri M, Aylin P. Systematic review of factors influencing length of stay in ICU after adult cardiac surgery. BMC Health Serv Res. 2016 Jul 29;16:318. doi: 10.1186/s12913-016-1591-3. PMID 27473872
- [Result] Tribuddharat S, Sathitkarnmanee T, Ngamsangsirisup K, Charuluxananan S, Hurst CP, Silarat S, Lertmemongkolchai G. Development of an open-heart intraoperative risk scoring model for predicting a prolonged intensive care unit stay. Biomed Res Int. 2014;2014:158051. doi: 10.1155/2014/158051. Epub 2014 Apr 10. PMID 24818129